CLINICAL TRIAL: NCT05362929
Title: Efficacy and Tolerability of a Hybrid Fractional Laser for the Treatment of Acne Scars in Patients With Skin of Color
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-14024
Record Dates: First submitted 2022-04-18; First posted 2022-05-05 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Acne Scars - Mixed Atrophic and Hypertrophic; Hyperpigmentation; Laser-Induced Hyperpigmentation
Keywords: skin of color; fitzpatrick skin type III; fitzpatrick skin type IV; fitzpatrick skin type V; acne scarring; sciton
MeSH Terms: conditions — Hypertrophy; Hyperpigmentation

STUDY DESIGN:
Intervention Model Description: This is a single-institution, baseline-controlled, prospective comparative study
Masking Description: Images of deidentified participants before and after treatment will be presented by two independent, non biased, blinded, board certified dermatologists for rating of improvement and outcome scores.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hybrid Fractional laser - SOC (Experimental): 23 participants with fitzpatrick skin type IV-V will be in this arm. At the first visit, participants will undergo informed consent, education about the procedure, education about proper sun-care, and will be provided sunscreen. Participants will be prescribed a prescription of hydroquinone or a retinol to prevent hyperpigmentation, per standard of care. If participants choose to take this they will wait one month of taking the prescription and then begin treatment sessions. If not, participants can begin treatment sessions right away. Treatment consists of 3 laser sessions with the Sciton Halo hybrid fractional laser. Session amount depends on the degree of improvement. At each session before and after images will be collected. At each session participants will fill out the dermatology quality of life survey as well as a patient satisfaction survey.
  Interventions: Device: Sciton Halo
- Hybrid Fractional laser- Non- SOC (Experimental): 23 participants with Fitzpatrick skin type I-III will be in this arm. At the first visit, participants will undergo informed consent, education about the procedure, education about proper sun-care, and will be provided sunscreen. Participants will be prescribed a prescription of hydroquinone or a retinol to prevent hyperpigmentation, per standard of care. If participants choose to take this they will wait one month of taking the prescription and then begin treatment sessions. If not, participants can begin treatment sessions right away. Treatment consists of 3 laser sessions with the Sciton Halo hybrid fractional laser. Session amount depends on the degree of improvement. At each session before and after images will be collected. At each session participants will fill out the dermatology quality of life survey as well as a patient satisfaction survey.
  Interventions: Device: Sciton Halo

INTERVENTIONS:
Device: Sciton Halo — Laser treatment
  Other Names: Sciton hybrid fractional laser; hybrid fractional laser; Serial number: 88086862

SUMMARY:
The investigators aim to investigate the efficacy and tolerability of a hybrid non-ablative/ablative laser for acne scarring in skin of color.

DETAILED DESCRIPTION:
Acne is chronic inflammatory condition involving the pilosebaceous unit. One of the most common complications of acne is scarring, which occurs as a result of dermal damage during the healing process of active acne. Studies have shown that acne scarring can have a negative impact on an individual's quality of life and has been described as a risk factor for multiple psychiatric conditions including depression, anxiety, suicide, and poor self-esteem. Unfortunately, treatment of acne scarring, particularly those of the atrophic subtype, prove difficult to treat. A 2016 Cochrane review failed to provide sufficient evidence to support the first-line use of any intervention. Laser technology has been emerging as an effective, non-invasive treatment of acne scarring. Ablative lasers work by delivering energy to the dermal layer of the skin, resulting in thermal injury and stimulation of dermal cells to produce collagen, thus resolving the scar. More recently, fractional lasers, which create multiple tiny columns of thermal injury, have been introduced with the benefit of reduced downtime and adverse effects compared to ablative lasers. The fractional CO2 laser is widely used for the treatment of acne scarring, however its use is limited in patients of Fitzpatrick IV and V skin due to risk of hyperpigmentation among other adverse events. The erbium-YAG fractional laser serves as an alternative, and has shown to produce less thermal injury and thus be more well-tolerated with lower risk of adverse effects in patients. The hybrid fractional laser combines a 2940 nm wavelength with a 1470 wavelength and has an ablative component targeting the epidermis and a nonablative component targeting the dermis at the same spot. The investigators seek to investigate the Sciton Halo, hybrid fractional laser for its efficacy in treating acne scarring and tolerability in patients with a specific emphasis on those with Fitzpatrick IV and V skin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females, ≥ 18 years of age at time of informed consent, seeking treatment for acne scarring
* Subject must voluntarily sign and date an IRB approved informed consent form
* Subjects with diagnosis of acne scarring recorded over the past 6 months
* Able to read, understand and voluntarily provide written informed consent.
* Subject is determined to be healthy, non-smoker
* Subjects able and willing to comply with the treatment protocol and follow-up schedule and requirements.
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period.

Exclusion Criteria:

* Subjects does not have the capacity to consent to the study
* subject underwent any acne scar treatments in the past 6 months prior to enrollment in the study
* Subject has active papulopustular or cystic acne within the past 6 months.
* Any history of keloidal scarring.
* Any previous surgical procedure in the treatment area in the past 12 months, or major surgery in the last 6 months.
* History of immunosuppression/immune deficiency disorders (including AIDS and HIV infection), and/or any history of systemic chemotherapy for prior 12 months.
* History or current use of the following prescription medications:

Immunosuppressive medications/biologics, 6 months prior to and during the study

* Accutane or other systemic retinoids within the past twelve months
* Smoking or vaping in the past 12 months.
* History of photosensitivity and/or connective tissue disease
* History of hyperlipidemia, diabetes mellitus, hepatitis, or bleeding disorders.
* History of major depressive disorders or endocrine disorders including but not limited to; hypothyroidism, Hashimoto's thyroiditis, or hyperthyroidism.
* History of ongoing pregnancy, active breastfeeding, cancer, and epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline acne scar severity | month 3
  2 Independent unbiased blinded dermatologists will rate before and after treatment images using Global Scale for Acne Scarring. This scale is rated on a scale of 0 to 5. 0 is the least severe, and 5 is the most severe.
Change from baseline acne scar severity | month 5
  2 Independent unbiased blinded dermatologists will rate before and after treatment images using Global Scale for Acne Scarring. This scale is rated on a scale of 0 to 5. 0 is the least severe, and 5 is the most severe.
Change from baseline acne scar severity | month 8
  2 Independent unbiased blinded dermatologists will rate before and after treatment images using Global Scale for Acne Scarring. This scale is rated on a scale of 0 to 5. 0 is the least severe, and 5 is the most severe.
Baseline Patient Satisfaction | month 0 (patient consultation visit )
  Patient Satisfaction Questionnaire. Questions are on a scale of -3 to 3, with -3 meaning the condition greatly decreased, and 3 meaning the condition greatly increased.
Patient Satisfaction | throughout study completion, an average of 8 months
  Patient Satisfaction Questionnaire. Questions are on a scale of -3 to 3, with -3 meaning the condition greatly decreased, and 3 meaning the condition greatly increased.
Patient Satisfaction | month 3
  Patient Satisfaction Questionnaire. Questions are on a scale of -3 to 3, with -3 meaning the condition greatly decreased, and 3 meaning the condition greatly increased.
Patient Satisfaction | month 5
  Patient Satisfaction Questionnaire. Questions are on a scale of -3 to 3, with -3 meaning the condition greatly decreased, and 3 meaning the condition greatly increased.
Patient Satisfaction | month 8
  Patient Satisfaction Questionnaire. Questions are on a scale of -3 to 3, with -3 meaning the condition greatly decreased, and 3 meaning the condition greatly increased.
Dermatology Quality of Life Survey Baseline | month 0 (patient consultation visit)
  Dermatology Life Quality Index. This is a standardized dermatology scale. Questions are subjectively answered by participants with answer choices ranging from "very much, a lot, a little, and not at all."
Dermatology Quality of Life Survey | throughout study completion, an average of 8 months
  Dermatology Life Quality Index. This is a standardized dermatology scale. Questions are subjectively answered by participants with answer choices ranging from "very much, a lot, a little, and not at all."
Dermatology Quality of Life Survey | month 3
  Dermatology Life Quality Index. This is a standardized dermatology scale. Questions are subjectively answered by participants with answer choices ranging from "very much, a lot, a little, and not at all."
Dermatology Quality of Life Survey | month 5
  Dermatology Life Quality Index. This is a standardized dermatology scale. Questions are subjectively answered by participants with answer choices ranging from "very much, a lot, a little, and not at all."
Dermatology Quality of Life Survey | month 8
  Dermatology Life Quality Index. This is a standardized dermatology scale. Questions are subjectively answered by participants with answer choices ranging from "very much, a lot, a little, and not at all."

CONTACTS AND LOCATIONS:
Overall Officials: Kseniya Kobets, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- 555 Taxter Road, Elmsford, New York, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will not be available to researchers not part of the original research team. All patient data will be de-identified.